CLINICAL TRIAL: NCT03878784
Title: Investigation of PACAP38-induced Headache and Rosacea-like Symptoms in Patients With Rosacea
Brief Title: PACAP38 Induced Headache and Rosacea-like Symptoms in Patients With Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Nita Katarina Frifelt Wienholtz, Principal Investigator, Medical Doctor, PhD Student, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RosMigExperiment
Record Dates: First submitted 2019-03-04; First posted 2019-03-18 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Sumatriptan; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACAP38 + Imigran (Active Comparator): Pituitary adenylate cyclase-activating peptide-38 infusion (10 picomol/kg/min) for 20 mins
  AND
  Imigrane infusion (0.4 mg/min) for 10 mins
  Interventions: Drug: Imigran
- PACAP38 + Isotonic Saline (Placebo Comparator): Pituitary adenylate cyclase-activating peptide-38 infusion (10 picomol/kg/min) for 20 mins
  AND
  Isotonic saline for 10 mins (placebo)
  Interventions: Other: Isotonic Saline

INTERVENTIONS:
Drug: Imigran — All patients will undergo this intervention on one of two study days
  Other Names: Sumatriptan
  Arms: PACAP38 + Imigran
Other: Isotonic Saline — All patients will undergo this intervention on one of two study days
  Arms: PACAP38 + Isotonic Saline

SUMMARY:
The investigators aim is to investigate the incidence of headache and rosacea-like flushing after pituitary adenylate cyclase-activating peptide-38 (PACAP38) with and without treatment with sumatriptan in patients with rosacea

DETAILED DESCRIPTION:
Pituitary adenylate cyclase-activating peptide-38 (PACAP38) plays a role in rosacea pathophysiology. Infusions of PACAP38 can trigger migraine-like attacks in migraine patients. PACAP38 also induces flushing which may imitate rosacea-like flushing. We are investigating whether the flushing after PACAP38 resembles rosacea-like flushing, and whether treatment with sumatriptan has an effect on the headache and flushing effects of PACAP38.

The purpose of this study is to investigate PACAP38-induced headache and flushing in patients with rosacea who have been treated with either sumatriptan or placebo using purpose-developed standardized interview. The investigators will use a double-blind, placebo-controlled crossover study design to investigate this.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with rosacea
* weight between 50 - 100 kilograms
* women in fertile age must not be pregnant and must use adequate contraception

Exclusion Criteria:

* migraine more than 5 days per month in average over the past year
* any primary headache other than migraine, apart from tension-type headache which must be less than 5 days per month
* headache < 48 hours before experimental day
* migraine < 72 hours before each experimental day
* daily / frequent use of any medication apart from contraceptive medication
* use of any drug less than 5 times the half-life of the drug at the time of the experiment
* women who are pregnant or breast-feeding at the time of the experiment
* anamnestic or clinical signs of hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) or hypotension (systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 50 mmHg)
* anamnestic or clinical signs of mental illness, or abuse of alcohol / drugs
* patients with glaucoma or prostate hyperplasia
* anamnestic or clinical symptoms of any sort that the investigating doctor deemed unfit for participating in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Incidence of headache and migraine | From 0 to 24 hours after infusion
  Incidence of PACAP38-induced headache and migraine-like attacks in patients with rosacea measured by numerical rating scale for pain from 0 ("no pain") to 10 ("worst pain imaginable") and international classification for migraine.
Effect of sumatriptan | From 0 to 24 hours after infusion
  Severity of PACAP38-induced headache after pretreatment with sumatriptan in rosacea patients measured by numerical rating scale for pain from 0 ("no pain") to 10 ("worst pain imaginable")

SECONDARY OUTCOMES:
Severity of flushing | From 0 to 4 hours after infusion
  Severity of PACAP38-induced flushing with and without sumatriptan-treatment measured by laser doppler flowmetry
Facial temperature | From 0 to 4 hours after infusion
  PACAP38-induced temperature changes with and without sumatriptan-treatment measured by infrared thermography
Superficial temporal artery diameter | From 0 to 4 hours after infusion
  Superficial temporal artery diameter after PACAP38 with and without sumatriptan-treatment measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD,PhD,DMSc, Principal Investigator — Professor
Locations (1):
- DanishHC, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wienholtz NKF, Christensen CE, Coskun H, Zhang DG, Ghanizada H, Egeberg A, Thyssen JP, Ashina M. Infusion of Pituitary Adenylate Cyclase-Activating Polypeptide-38 in Patients with Rosacea Induces Flushing and Facial Edema that Can Be Attenuated by Sumatriptan. J Invest Dermatol. 2021 Jul;141(7):1687-1698. doi: 10.1016/j.jid.2021.02.002. Epub 2021 Feb 16. PMID 33600826